CLINICAL TRIAL: NCT06150937
Title: HIV Self-testing Intervention for Female Sex Workers Who Inject Drugs in Kazakhstan
Brief Title: HST for Female Sex Workers/Drug Users in Kazakhstan
Acronym: AEGIDA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Victoria Frye, Medical Professor, City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34DA049664 (NIH)
Record Dates: First submitted 2023-11-14; First posted 2023-11-30 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: HIV Testing; Intention
Keywords: Pre-exposure Prophylaxis; Post-exposure Prophylaxis; HIV self-testing

STUDY DESIGN:
Intervention Model Description: Pilot RCT of a 4-session intervention. Participants will be randomized in a 2:1 intervention to control ratio and followed up for 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AEGIDA intervention arm (Experimental): Four session behavioral intervention to promote consistent HIV testing, frequent HIV testing and intention to uptake PEP/PrEP.
  Interventions: Behavioral: AEGIDA intervention arm
- AEGIDA control arm (Active Comparator): Four session didactic intervention to promote self-screening for common health problems, including HIV self-testing.
  Interventions: Behavioral: AEGIDA control arm

INTERVENTIONS:
Behavioral: AEGIDA intervention arm — The intervention arm has 4 sessions facilitated one-on-one by trained staff and lasting ~40 minutes. The first session focuses on establishing rapport, assessing HIV risk, and educating/training participants on HIV self-testing/PEP/PrEP. The second session on peer education/training, barriers to and facilitators of testing, and supporting peers in receiving reactive and/or indeterminate HIV test results, as well as self-care. The third session on stigma and discrimination and techniques to cope with and resist stigma. The final session is a culminating one focused on reviewing key skills and health promotion planning conducted in first three sessions. The intervention arm applies anti-intersectional stigma, empowerment, and harm reduction approaches. All participants will receive/have access to HIV self-test kits every three months.
  Arms: AEGIDA intervention arm
Behavioral: AEGIDA control arm — The control arm has 4 sessions via one-on-one facilitation by a trained facilitator and lasting ~40 minutes. It includes basic information on self-screening for common adverse health conditions among women in Kazakhstan, including STIs and HIV, as well as information on testing and risk reduction. All participants will receive/have access to HIV self-test kits every three months.
  Arms: AEGIDA control arm

SUMMARY:
The goal of this behavioral intervention clinical trial is to assess acceptability, feasibility, and preliminary efficacy of a 4-session intervention to increase consistent HIV testing and linkage to care and prevention among HIV uninfected (assessed via on-site testing) female sex workers who use drugs in Kazakhstan.

The main question it aims to answer are:

1. is the intervention acceptable and feasible
2. do participants randomized to the intervention arm report: 1) past 3-month testing; 2) frequent testing (2+ test over 6 mos.); 3) linkage to HIV care and ART initiation, if positive, or intention to uptake PrEP, if negative, as compared with control arm participants. Secondary outcomes include incident, biologically-confirmed STIs and stigma-related factors. Follow-up period is six months.

All participants will be HIV-negative upon study enrollment as assessed via rapid HIV test.

Participants randomized to the intervention arm will be engaged in a 4-session intervention that offers training and education in HIV self-testing, peer education on HIV self-testing, internalized stigma coping and resistance via basic cognitive restructuring, and provision of HIV self-test kits and reminders every three months. Researchers will compare participants randomized to the intervention arm to participants randomized to the time- and attention-control arm to evaluate impact of the intervention on the outcomes described above.

DETAILED DESCRIPTION:
SPECIFIC AIMS This application seeks to transfer R34 DA049664, awarded previously to Research Foundation City University of New York (Contact MPI: Frye), to Columbia University where both the Contact and non-Contact MPI (El-Bassel) are based. The goal of this study is to assess acceptability, feasibility, and preliminary efficacy of an intervention to increase consistent HIV testing and linkage to care and prevention among female sex workers who inject drugs (FSWID) in Kazakhstan. Central Asia (CA) has one of the world's fastest growing HIV epidemics, increasing 30% since 20101. Key populations made up 95% of new infections in 2017, with 9% among female sex workers (FSW), 39% among people who inject drugs (PWID), and 28% among clients/sex partners of key populations. In Kazakhstan, new HIV infections doubled from 2010 to 2017 and AIDS-related deaths increased 32%. According to the Kazakh Scientific Center of Dermatology and Infectious Diseases (KSCDID), HIV prevalence is 9% among PWID and 2% among FSW, and incidence increased among both groups from 2016 to 2017. Overall, 79% of people living with HIV (PLWH) were status aware, 43% on antiretroviral therapy (ART), and 24% virally suppressed in 2017. FSW who inject drugs (FSWID) are at increased risk of HIV/STI infection and less likely to test/receive care. Prior research found that ~30% of FSWID are HIV-infected.

HIV testing is the point of entry to HIV care and prevention, including PrEP/PEP where available. Consistent testing and early diagnosis are essential to achieving global 90-90-90 targets (90% status aware; 90% on ART; 90% virally suppressed). HIV-related stigmas, including community, enacted/experienced, internalized/self- and anticipated, remain major barriers to HIV testing, care and prevention. FSWID in Kazakhstan experience dual stigma and bias from healthcare providers (HCPs) related to sex work and/or drug use. HIV self-testing (HST) is an acceptable, user-controlled tool that increases new case identification and, due to less contact with HCPs, reduces enacted and anticipated stigma. HST interventions for FSW in Africa increased status knowledge, recent testing and HST is WHO recommended for key populations although reading test results and suboptimal linkage to care are concerns. There is a tension between HST as a private, stigma-avoidant approach and linkage to care/prevention, which is face-to-face. Prior research suggests that FSW welcome HST, but that HCP bias inhibits linkage to care. As PrEP may become available for key populations in CA, interventions to leverage HST to locate new cases via consistent testing and facilitate ART and biomedical prevention linkage are needed. Presently, no such interventions are registered or have been evaluated for FSWID in CA. To address this gap, the study proposes to design and assess feasibility, acceptability and preliminary efficacy of a novel, theory-based intervention for FSWID that will combine core components from efficacious HST and linkage interventions with novel components to reduce self-stigma and improve anticipated stigma coping, as well as exploratory targets (e.g. HCP/community stigma, collective efficacy, PrEP awareness/intention, etc.) identified via formative research. Finally, the study will describe data required to calculate cost implications related to feasibility/sustainability. The study aims are:

Aim 1: Elicit preferences to inform adaptation of existing evidence-based HST components: training (peer vs. pro), distribution (network vs. site), support (in-person vs. text) and linkage (navigation, etc.). Elicit perspectives to inform design of novel linkage to care/biomedical prevention components. To achieve this aim, the following will occur: formative research (30 in-depth interviews; 4 focus groups [N=20]) to identify preferences around HST; and characterize barriers (e.g. HCP/community/anticipated stigma/self-stigma) to and facilitators of (e.g. self and collective efficacy, empowerment, peer support, PrEP awareness) linkage to care/prevention.

Aim 2. Design, component test (N=20) and pre-pilot (N=20) the 4-session intervention. Here, modified intervention adaptation and design will be used to combine core components of efficacious HST interventions for FSW with novel ones to address self-stigma and anticipated stigma coping, as well as advocacy and peer-based linkage facilitators, using stigma, advocacy, and empowerment theoretical approaches.

Aim 3. Aim 3. Assess feasibility, acceptability, and preliminary efficacy of the intervention in increasing HIV testing and linkage to care (if positive) or biomedical uptake intention (if negative). To achieve this aim, the study will randomize 90 HIV-negative FSWID to a 4-session experimental arm or a time- and attention-controlled standard HIV test/risk reduction counseling arm and follow them for 6 months. Primary outcomes are: 1) past 3-month testing; 2) frequent testing (2+ test over 6 mos.); 3) linkage to HIV care and ART initiation, if positive; and 3) intention to uptake PrEP if negative. Secondary outcomes will include incident, biologically-confirmed STIs and stigma-related factors.

The pilot RCT will be conducted in partnership with Amelia, a non-profit, FSW advocacy organization, and KSCDID, which leads national HIV treatment/prevention strategy. The study builds on GHRCCA's decade-long success in designing and testing HIV behavior change interventions in Kazakhstan, significant regional research infrastructure, providing economies in execution. The results of this study, which is unique in linking HST with stigma-reduction approaches, will inform the submission of an R01 application and will have implications for research with FSW and PWID globally and in the United States.

ELIGIBILITY:
Inclusion Criteria:

* report vaginal or anal intercourse in past year in exchange for money, alcohol, drugs, or other goods/resources
* report having injected or used drugs and/or binged alcohol in past year
* report at least one episode of condomless sexual intercourse in past 90 days with a paying, casual, or regular (intimate) sexual partner
* HIV-negative as confirmed by rapid test at enrollment

Exclusion Criteria:

* have a cognitive or psychiatric impairment preventing comprehension of study procedures as assessed during Informed Consent
* do not speak and understand Russian at a conversational level
* previously enrolled in the pre-pilot portion of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
HIV testing | 6 months
  HIV testing (operationalized as 1+ test in past 3 mos. over follow-up) When was the last time you were tested for HIV? (6M_HIV TEST LAST)
  1. In the past 3 months
  2. Not in the past 3 months, but in the past 6 months
  3. Not in the past 6 months, but in the past year
  4. Not in the past year, but in the past 3 years
  5. More than 3 years ago
  99. Refuse to answer
Frequent HIV testing | 6 months
  frequent HIV testing (2+ test within 6 mos. over follow-up) In the last 3 months, how many times have you tested for HIV? (6M_HIV TEST TIMES) 0 (never)
  1. time
  2. times 3-4 times
  5 or more times
HIV care linkage/ART initiation | 6 months
  self-reported HIV care receipt and ART initiation For participant's who test positive, the study team engages in outreach and linkage to care, which is documented in the study file
Intention to uptake PrEP | 6 months
  self-reported intention to use PrEP Have you heard of "PrEP" also known as pre exposure prophylaxis?
  In the last three months, have you spoken to a health care provider about PrEP to reduce the risk of HIV infection?
  In the last three months, have you taken PrEP to reduce the risk of HIV infection?
  Are you currently taking PrEP (pre-exposure prophylaxis)?
  Are you taking PrEP under a doctor or health care professional's supervision?
  Are you planning to take PrEP (pre-exposure prophylaxis)?
  Women who exchange sex and/or use drugs should take PrEP.
  Based on what I know about PrEP, I would prefer (RANK the options):

SECONDARY OUTCOMES:
incident STI | 12 months
  incident, biologically-confirmed STIs
stigma-related outcomes | 12 months
  self-reported internalized HIV stigma, sex worker stigma, drug user stigma
  Smith LR, Earnshaw VA, Copenhaver MM, Cunningham CO. Substance use stigma: Reliability and validity of a theory-based scale for substance-using populations. Drug Alcohol Depend. 2016 May 1;162:34-43. doi: 10.1016/j.drugalcdep.2016.02.019. Epub 2016 Feb 26. PMID: 26972790; PMCID: PMC5293183.
  Kerrigan, D., Karver, T., Barrington, C., Davis, D. A., Donastorg, Y., Perez, M., . . . Chan, K. S.
  (2021). Using Item Response Theory to Develop the Experiences of Sex Work Stigma Scale: Implications for the Reseaerch on the Social Determinants of HIV. AIDS Behavior.
  With the new HIV medications, HIV infection is no longer a danger. (6M HIV KNOW MED). (G04) True False Don't know

CONTACTS AND LOCATIONS:
Locations (1):
- Global Health Research Center of Central Asia, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] West BS, Darisheva M, McCrimmon T, Chang M, Zholnerova N, Grigorchuk E, Starbird L, Terlikbayeva A, Primbetova S, Cordingley O, Baiserkin B, Kassymbekova S, Mussina Z, Rashidov I, Gilbert L, El-Bassel N, Frye V; AEGIDA Study Team; Key Community Partners. AEGIDA: Results of a Pilot Randomized Trial of an HIV Self-Testing Intervention for Women Who Exchange Sex and Use Substances in Kazakhstan. AIDS Behav. 2025 Nov 3. doi: 10.1007/s10461-025-04927-0. Online ahead of print. PMID 41177842